CLINICAL TRIAL: NCT05616351
Title: Antibiotische Therapie In Infektionen Des Diabetischen Fusssyndroms
Brief Title: Antibiotic Therapy in Infections of the Diabetic Foot Syndrome
Acronym: DFO
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01512; mu22Mueller2
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Foot Infection
Keywords: diabetic foot syndrome; antibiotic therapy; soft tissue infection; osteomyelitis; bone infection
MeSH Terms: conditions — Soft Tissue Infections; Osteomyelitis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection in patients with diabetic foot syndrome and infections in the area of the foot — Data collection: on (surgical and antibiotic) treatment and implementation of the recommendations published 2019 with regard to the duration of antibiotic therapy.

SUMMARY:
This retrospective study examines the surgical and antibiotic treatment of diabetic foot syndrome infections treated at the University Hospital Basel since 2019.

It analyses the implementation of the hospital in-house guidelines published in 2019 with regard to antibiotic therapy in diabetic foot infections, taking into account clinical, microbiological and histopathological criteria. The defined endpoints are (i) fully compliant with internal policies, (ii) partially compliant with internal policies, and (iii) not compliant with internal policies. The recording of these proportions is descriptive.

DETAILED DESCRIPTION:
This retrospective study examines the surgical and antibiotic treatment of diabetic foot syndrome infections treated at the University Hospital Basel since 2019. (In 2019 the departments of infectiology and orthopedics at the University Hospital Basel published recommendations with regard to the duration of antibiotic therapy in infections of the diabetic foot syndrome. This depends on whether a surgical intervention was performed and takes into account both the microbiological and the histopathological samples). Data that are routinely collected in everyday clinical practice and stored in the hospitals' medical records will be evaluated. The aim of this research project is to check the implementation of these recommendations.

Inadequate use of antibiotics should thus be recognized. The study has the aspect of quality control.

ELIGIBILITY:
Inclusion Criteria:

* soft tissue infection or bone infection (incl. osteomyelitis) in diabetic foot syndrome
* inpatient stay at the University Hospital Basel between January 1st, 2019 and December 31st, 2021
* surgical intervention (amputation and/or debridement)
* signed general consent

Exclusion Criteria:

* datasets without a diagnosis of the diabetic foot
* no surgical intervention performed (amputation and/or debridement)
* surgical interventions performed by disciplines other than orthopaedics/traumatology (e.g. vascular surgery)
* infections in osteosynthesis material (implant or fracture-associated infections)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data in this retrospective study derive from everyday clinical work, collected between January 1st, 2019 and December 31st, 2021 at the Department of Infectiology and Department of Orthopaedics and Traumatology at the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Compliance with the hospital in-house guidelines for diabetic foot infections with regard to antibiotic treatment | one time assessment at baseline
  Implementation of the guidelines published in 2019 with regard to antibiotic therapy in diabetic foot infections, taking into account clinical, microbiological and histopathological criteria. The defined endpoints are (i) fully compliant with internal policies, (ii) partially compliant with internal policies, and (iii) not compliant with internal policies.

SECONDARY OUTCOMES:
Duration of antibiotic therapy (days) | one time assessment at baseline
  Duration of antibiotic therapy
Relapse of diabetic foot infections (number) | one time assessment at baseline
  Relapse of diabetic foot infections (number)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Marc Müller, Prof. Dr. med., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- University Hospital Basel, Orthopedics and Traumatology, Basel, Switzerland

REFERENCES:
- [Result] Reinert N, Wetzel K, Franzeck F, Morgenstern M, Aschwanden M, Wolff T, Clauss M, Sendi P. What is the agreement between principles and practice of antibiotic stewardship in the management of diabetic foot infection: an in-hospital quality control study. J Bone Jt Infect. 2024 Jun 28;9(3):183-190. doi: 10.5194/jbji-9-183-2024. eCollection 2024. PMID 39040989
- See also: Link to citation — https://jbji.copernicus.org/articles/9/183/2024/jbji-9-183-2024.pdf